CLINICAL TRIAL: NCT03631836
Title: Phase I Study of Monoclonal Antibondy (GS) 5745, an Matix Metalloproteinase 9 (MMP9) Mab Inhibitor, in Combination With Bevacizumab in Patients With Recurrent Glioblastoma
Acronym: MARELLE01
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-65
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Antibodies, Monoclonal; Bevacizumab; Blood Specimen Collection; Dynamic Contrast Enhanced Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combinaton monoclonal therapeutic antibody and bevacizumab (Experimental): Determine the safety profile and tolerability of monoclonal therapeutic antibody given in combination with a fixed dose of bevacizumab in patients with recurrent glioblastoma in terms of Dose-Limiting Toxicities
  Interventions: Drug: Monoclonal antibody; Drug: Bevacizumab; Biological: Blood sample; Device: Dynamic Contrast Enhanced magnetic resonance imaging (DCE-MRI)

INTERVENTIONS:
Drug: Monoclonal antibody — 3 doses of Monoclonal antibody could be tested
Drug: Bevacizumab — fixed dose of bevacizumab (10 mg/ kg every two weeks)
Biological: Blood sample — Evaluate the biomarkers plasma levels during administration of drug
Device: Dynamic Contrast Enhanced magnetic resonance imaging (DCE-MRI) — Assess antiangiogenic effects by DCE-MRI

SUMMARY:
Despite surgery and first-line standard of care which consist of radiotherapy with concomitant and adjuvant temozolomide, all patients with glioblastoma (GB) will experience relapse. At the time of recurrence, therapeutic options include surgery or reirradiation in selected cases, while in other cases, bevacizumab, approved by Food and Drug Administration (FDA) but not European Medicines Agency (EMA), is the preferred option worldwide. Primary and acquired resistance to bevacizumab has been explored without definitive finding.

Biomarkers able to predict response to antiangiogenic agents and particularly to bevacizumab are an unmet medical need. We have showed that a low Matrix metallopeptidase 9 (MMP9) or a high Matrix metallopeptidase 2 (MMP2) baseline plasma levels were associated with a high response rate and a prolonged Progression-free survival (PFS) and overall survival (OS) in recurrent GB patients treated with bevacizumab but not with cytotoxic chemotherapy. We also observed that MMP9 plasma level decreased during bevacizumab treatment and tend to increase at progression. Finally, in a retrospective analysis performed in the Avaglio trial (a randomized phase III trial that tested bevacizumab versus placebo in addition to standard of care in patients with newly diagnosed glioblastoma), a low plasma level of MMP9 at baseline predicted consistently PFS and OS gain associated to bevacizumab.

These results are consistent with the role of MMP9 in vasculogenesis, since MMP9 contribute to the recruitment of circulating endothelial and myeloid precursors, an alternative vascularization process which is in part independent of the vascular endothelial growth factor (VEGF) pathway.

Monoclonal Antibody (GS) 5745 is specifically directed against MMP9. First in human phase I study has been completed. Development is ongoing.

Our results strongly support a role for MMP9 in the primary or acquired resistance to bevacizumab. Therefore, we hypothesize that the Monoclonal Antibody GS5745 may overcome resistance to bevacizumab through a specific inhibition of MMP9. While a preclinical program is initiated in our lab, the proposed phase I study is the first step to analyze the tolerance, determine the recommended dose of the combination and explore the impact of GS5745 on MMP9 plasma levels and multimodal imaging in patients with recurrent glioblastoma.

Objective:

Determine the safety profile and tolerability of GS5745 given in combination with a fixed dose of bevacizumab in patients with recurrent GB in terms of Dose-Limiting Toxicities.

Multicenter, open label, dose-finding study of GS5745 in combination with bevacizumab administered at a fixed dose; both drugs will be administered once every two weeks for a total treatment duration of a maximum of 12 months.

Before initiation of each new dose level, a meeting between the sponsor, the coordinator, the investigators and an independent external expert will take place to decide jointly the next dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of isocitrate dehydrogenase (IDH) wild-type glioblastoma
* First or second recurrence after standard treatment with combined chemo-irradiation
* Patients must have measurable tumour disease as defined by Response assessment in neuro-oncology (RANO) criteria within 2 weeks before the first drug administration
* Stable or decreasing dose of corticosteroids within 5 days prior first administration
* Karnofsky Performance Status superior at 60%
* Negative serum or urine pregnancy test done inferior or egal at 7 days prior to registration, for women of childbearing potential only
* Provide informed written consent

Exclusion Criteria:

* Major surgery (including craniotomy) within 4 weeks prior to the first day of study drug administration
* Chemotherapy within 4 weeks prior to the first day of study drug administration
* Radiotherapy within 3 months prior the diagnosis of progression.
* Prior treatment with bevacizumab or other vascular endothelial growth factor (VEGF) receptor targeted agent
* Evidence of Central Nervous System (CNS) haemorrhage on the baseline MRI.
* Other conditions reported to exclude bevacizumab administration
* Men or women of childbearing potential who are unwilling to employ adequate contraception during this study
* Concomitant serious immunocompromised status
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy within 5 years of registration. Exceptions: Non-melanotic skin cancer or carcinoma-in-situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Determine the Dose Limiting Toxicity (DLT) | 36 months
  Toxicities are to be graded according to the Common Terminology Criteria for Adverse Events (CTCAE). Any grade 4 event and selected grade 3 events of any duration.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Director, Study Director — Assistance Publique des Hôpitaux de Marseille
Locations (1):
- Assistance Publique des Hôpitaux de Marseille, Marseille, France